CLINICAL TRIAL: NCT03857087
Title: Gallium-68 Prostate Specific Membrane Antigen for Ovarian Cancer: A Pilot Feasibility Study
Brief Title: 68Ga-PSMA PET in Diagnosing Metastasis in Patients With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Principal Investigator, Michael Ohliger, MD, Assistant Professor, University of California, San Francisco
Other Study IDs: 174017; NCI-2018-02331 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnostic 68Ga PSMA PET/MRI: Patients receive gallium Ga 68-labeled PSMA-11 IV over 1-2 minutes. After about 60 minutes, patients undergo PET/MRI for approximately over 50-60 minutes. Patients may undergo an optional repeat gallium Ga 68-labeled PSMA-11 PET between 8 and 12 weeks after completion of the first PET/MRI.
  Interventions: Drug: Gallium Ga 68-labeled PSMA-11; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: Gallium Ga 68-labeled PSMA-11 — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA-11; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; PSMA-HBED-CC GA-68
Procedure: Magnetic Resonance Imaging (MRI) — Given PET/MRI
  Other Names: Magnetic Resonance Imaging; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging (NMRI)
Procedure: Positron Emission Tomography (PET) — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies how well gallium Ga 68-labeled prostate specific membrane antigen (PSMA)-11 (68Ga-PSMA) positron emission tomography (PET) works in patients with ovarian cancer to detect whether the tumor has spread to other places in the body. 68Ga-PSMA is a radioactive substance that binds to blood vessels around the ovarian cancer and can be imaged using PET. Diagnostic procedures, such as PET, may help find and diagnose find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and utility of 68Ga-PSMA PET imaging patients with ovarian cancer.

II. Determine detection sensitivity for nodal metastases for PSMA PET stratified by node size.

SECONDARY OBJECTIVES:

I. To assess the correlation between targeted molecular uptake of 68Ga-PSMA PET and PSMA expression in surgical resection specimens.

EXPLORATORY OBJECTIVES:

I. To explore heterogeneity of 68Ga-PSMA PET uptake in cases of metastatic ovarian cancer.

II. To determine the relationship between 68Ga-PSMA PET uptake, diffusion weighted imaging, and MRI-derived tumor perfusion.

OUTLINE:

Patients receive gallium Ga 68-labeled PSMA-11 intravenously (IV) over 1-2 minutes. After about 60 minutes, patients undergo PET/magnetic resonance imaging (MRI) for approximately over 50-60 minutes. Patients may undergo an optional repeat gallium Ga 68-labeled PSMA-11 PET between 8 and 12 weeks after completion of the first PET/MRI.

After completion of study, patients are followed up at 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with one of the following, identified on prior imaging (CT, MRI or Ultrasound):

   1. adnexal mass
   2. abdominal or pelvic tumor suspicious for ovarian cancer metastases (either suspected on clinical grounds, or known from prior tissue sampling)
2. Female,
3. Age >= 18 years
4. Creatinine </= 1.5 mg/dL
5. Ability to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Patient unlikely to comply with study procedure, restrictions and requirements and judged by the investigator to be unsuitable for study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will be women with adnexal masses or other lesions suspicious for ovarian cancer metastases, who are scheduled for either resection or chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of gallium Ga 68-labeled PSMA-11 positron emission tomography (PET) positive lesions detected by standard staging scans | Study Visit Day 1
  Will be descriptively reported for each patient and correlated with the lesions observed in standard imaging computed tomography/magnetic resonance imaging (CT/MRI). In addition, the mean, range, and standard deviation of standardized uptake value maximum (SUVmax) (across all visualized lesions per patient) and SUVmax-average (ave) (across all patients in the study cohort) will be descriptively reported.
Number of overall ovarian cancer lesions detected by standard staging scans | Study Visit Day 1
  Will be descriptively reported for each patient and correlated with the lesions observed in standard imaging CT/MRI.
Average maximum standard uptake value (SUVmax) | Study Visit Day 1
  The mean, range, and standard deviation of SUVmax across all visualized lesions per patient will be descriptively reported.
Number of lymph nodes detected by PET | Study Visit Day 1
  Will be compared and stratified by lymph node size. For patients undergoing surgical resection, this will be compared with the number of involved lymph nodes by surgical resection. For lymph nodes that are not resected, the behavior on follow-up clinical CT scans (if available) will be used to assess for involvement.
Number of lymph nodes detected by MRI | Study Visit Day 1
  Will be compared and stratified by lymph node size. For patients undergoing surgical resection, this will be compared with the number of involved lymph nodes by surgical resection. For lymph nodes that are not resected, the behavior on follow-up clinical CT scans (if available) will be used to assess for involvement.

SECONDARY OUTCOMES:
Correlation between targeted molecular uptake of 68Ga-PSMA PET and prostate-specific membrane antigen (PSMA) expression in surgical resection specimens | Study Visit Day 1
  For patients undergoing surgical resection, the 68Ga PSMA-PET uptake will be correlated with PSMA expression in the primary tumor as well as metastatic sites. PSMA expression measurement is available as a core service from the cancer center

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ohliger, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kunikowska J, Bizon M, Pelka K, Derlatka P, Olszewski M, Krolicki L. 68 Ga-Prostate-Specific Membrane Antigen PET/CT in Ovarian Tumors : Potential to Differentiate Benign and Malignant Tumors Before Surgery: A Preliminary Report. Clin Nucl Med. 2023 Feb 1;48(2):e60-e66. doi: 10.1097/RLU.0000000000004486. Epub 2022 Nov 18. PMID 36512649